CLINICAL TRIAL: NCT06916533
Title: Effectiveness of ENBORTH-TR Intervention on Pain, Quality of Life, Sleep Quality, Kinesiophobia, Perceived Occupational Performance and Satisfaction in Low Back and/or Neck Pain: A Single Blind Randomised Controlled Study
Brief Title: ENBORTH-TR Intervention for Back/Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Berkan Torpil, PhD, Assoc Prof, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/209
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-03

CONDITIONS: Low Back Pain; Neck Pain
Keywords: low back pain; neck pain; quality of life; sleep quality; occupational performance; satisfaction; kinesiophobia
MeSH Terms: conditions — Low Back Pain; Neck Pain; Sleep Initiation and Maintenance Disorders; Personal Satisfaction; Kinesiophobia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Experimental): According to the evaluation results, client-centred occupational therapy intervention was applied to this group. The client-centred occupational therapy intervention is based on the activities that the participants stated in the COPM in the first evaluation and had problems.
  Interventions: Behavioral: Client-centred Occupational Therapy Intervention Group
- ENBORTH-TR Invertention Group (Experimental): In this study, ENBORTH-TR training programme is applied in addition to person-centred intervention. ENBORTH-TR programme starts from the definition of pain, explains its mechanism, affected muscle groups, and provides awareness training that will improve the quality of life of individuals in pain management such as environmental regulations, relaxation techniques, stress management.
  Interventions: Behavioral: ENBORTH-TR Intervention; Behavioral: Client-centred Occupational Therapy Intervention Group

INTERVENTIONS:
Behavioral: ENBORTH-TR Intervention — This intervention program is structured with a multifaceted and holistic approach, starting with the definition of pain and covering topics such as basic body anatomy, functions and pain mechanisms, ergonomics training, environmental regulations, psychosocial factors such as stress, relaxation techniques, sleep and time management.
  Arms: ENBORTH-TR Invertention Group
Behavioral: Client-centred Occupational Therapy Intervention Group — Client-centered occupational therapy intervention consists of 5 stages: (1) Client-centered goal setting, (2) creation of the therapy plan, (3) implementation of interventions, (4) evaluation of results, and (5) obtaining feedback.

SUMMARY:
This study was conducted to investigate the effectiveness of the ENBORTH-TR training programme given in addition to client-centred intervention in individuals with low back and/or neck pain. The current study investigates the effect of ENBORTH-TR on pain, quality of life, sleep quality, kinesiophobia and perceived occupational performance and satisfaction levels. This study was designed according to the CONSORT statement, which provides standardisation in randomised controlled trials. In addition, the study was approved by the scientific research ethics committee of a university. Written informed consent was obtained from all participants before the study.

DETAILED DESCRIPTION:
This study was planned as a single-blind randomized controlled trial and was conducted using the CONSORT checklist. Participants who met the inclusion and exclusion criteria and signed the written consent form were divided into 2 groups by simple randomization. While the client-centered intervention procedure was applied to both groups within the scope of the study, the ENBORTH-TR intervention procedure was also applied to the intervention group. All intervention procedures in the study were planned with the telerehabilitation method for 3 days a week for 4 weeks and each session was planned to consist of 45-minute sessions. A total of 136 people were included in the study, 69 in the control group and 67 in the intervention group.

Interventions Client-centered intervention procedure

Using the literature, a client-centered intervention procedure for individuals with low back and/or neck pain was developed. This intervention procedure consists of 5 steps. These steps are as follows:

First phase: Setting measurable, realistic and achievable goals to address occupational performance issues

Second phase: Developing and evaluating the pros and cons of possible solutions by brainstorming on the oupations identified by the Canadian Occupational Performance Measure.

Third stage: Deciding on a solution, making a plan and implementing it. At this stage, adaptations are made to the oupations with problems, a new oupation is chosen and the oupation is prioritized.

Fourth stage Reviewing the results of the client-centered intervention process

Fifth stage: Receiving feedback on the individual's experiences and making changes where necessary.

Client-centered intervention is known as a core component, a historically integrated value and a fundamental element of occupational therapy interventions. It is based on focusing on the individual's values, needs and goals by prioritizing the individuals' own experiences and preferences. Within the scope of the intervention procedure, telerehabilitation method was applied jointly to both groups. In the first evaluations, occupational performance problems were identified according to the Canadian Occupational Performance Measure data. The participants were given a general information about the problem areas and the intervention process and the session contents were planned. In the sessions, it was aimed to step, prioritize, analyze and break down the occupations for low back and/or neck pain, apply specific interventions to the areas of difficulty and adapt the occupation according to individual needs when necessary. Within the framework of a holistic approach, it was aimed to evaluate environmental and psychosocial factors and to identify and support areas that can be intervened.

ENBORTH-TR intervention:

This training program was given to the intervention group in addition to the client-centered intervention. This intervention, which was carried out with the telerehabilitation method, continued for a total of 4 weeks, 3 days a week and 45-minute sessions. The program consists of 5 stages and the content of the training is discussed in detail below. In order to make the program more understandable, the training was carried out with a booklet supported by videos and visuals. The name of the intervention program consists of the initials of the words "Ergoteraphy, Neck, Back, Orthopaedics". This intervention was created by utilizing the literature. The contents of the 5 stages of the intervention are presented below:

Stage 1: Basic Information: Body anatomy, Functions and Pain Mechanisms:

This phase covers sessions 1-3. The main purpose of the sessions is to enable the clients to recognize their bodies and the pain they experience, to gain awareness, to establish a relationship of trust between the therapist and the client and to set goals.

Stage 2: Ergonomics Training and Environmental Arrangements:

In sessions 4-6, clients' living spaces were evaluated and ergonomic adjustments were made for low back and/or neck pain. In addition to these adjustments, joint and energy conservation techniques were taught and information was given about correct movement patterns and body mechanics.

Stage 3: Psychosocial Factors, Sleep and Time Management:

Sessions 7 and 8 focused on psychosocial factors and sleep. Progressive muscle relaxation technique was taught and practiced and sleep diary application was explained. In addition, pre-sleep nutrition and sleep habits were emphasized. Sessions 9 and 10 focused on time management. Time management aims not only to increase productivity, but also to reduce pain, conserve energy and manage stress, thus supporting the individual's participation and quality of life.

Stage 4: Client Feedback At this stage, the extent to which the clients were able to transfer the information learned in the training to daily life was evaluated. At the same time, the training process was also reviewed in general, and areas that were missing or needed to be reinforced were identified. Thus, it was aimed to complete the training in a healthy way

Stage 5: Revisiting Feedback In the last stage, according to the feedback received from the clients, the areas that were not understood or thought to be missing were reconsidered. The training process was completed by answering the questions posed by the clients regarding the training process and the readings.

Statistically analysis Data were analyzed with SPSS version 27.0 statistical software package program. The normality of the data was analyzed by using Kolmogorov-Smirnov test. Nonparametric tests were used because the data did not show a normal distribution. Differences between groups were analyzed with chi-square test for nominal data. Comparisons between the groups were conducted by using the Mann-Whitney U test. Pre- to post-intervention changes within the groups were analyzed with the Wilcoxon signed-rank test. Significance was evaluated at levels of 0.05. Effect size was calculated by using the means and standard deviations of the groups. Effect size benchmarks were determined as <0.30, 0.30-0.80, and >0.80 and considered small, moderate, and strong, respectively.

ELIGIBILITY:
Inclusion Criteria:

* To be at least primary school graduate
* Participating in the study voluntarily
* To be able to read and write Turkish
* At least 24 points from the Mini Mental State Examination
* Having low back and neck pain for 3 months or more
* Being between the ages of 18-65

Exclusion Criteria:

1. Having a neurological, psychiatric or chronic disease (cancer, etc.) or having any secondary disease that will adversely affect the work
2. History of any malignancy or spinal fracture
3. Having undergone a surgical procedure for low back and/or neck pain or having undergone any other surgical intervention within the last 6 months
4. Not participating regularly in the intervention process
5. Participating in another rehabilitation program during the study period

7) Diagnosis of pregnancy or suspected pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 136 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-04-05 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | 30 minutes
  COPM, which is most frequently used among occupational therapists, is a standardised measurement tool used to determine the individual's activity performance problems and to measure performance satisfaction. In the COPM, which is a semi-structured interview, individuals evaluate their activity preferences with performance and satisfaction scores given by themselves. Individuals are asked about their activity performance problems and concerns about 3 areas including self-care, productivity and leisure time activities. Up to three problems can be identified in each activity area (self-care, productivity, leisure). Performance and satisfaction scores are again determined by the individual between 1 and 10 points.
Visual Analog Scale (VAS) | 5 minutes
  Visual analogue scale was used to assess the pain intensity of the participants. During the assessment, the participants were asked to mark the points where they felt pain during sleep, rest and activity on a 10 cm horizontal line with the left end 0 meaning 'no pain' and the right end 10 meaning 'very severe pain'. Before marking, the individuals were explained in detail what they should do. Then, the distance of the marked points to point 0 was measured and recorded in centimetres
Tampa Scale of Kinesiophobia (TSK) | 7 minutes
  The TSK, which is used in the evaluation of kinesiophobia, is a Likert-type scale consisting of 17 questions. Each question is scored between 1 and 4 points (1 = strongly disagree to 4 = strongly agree). The lowest score that can be obtained from the scale is 17 and the highest score is 68. A high score in the total score of the scale indicates a high level of kinesiophobia.
Nottingham Health Profile (NHP) | 10 minutes
  The NHP used to assess the people's QoL consists of a total of 38 questions. It has 6 subscales and assesses energy, pain, emotional reactions, sleep, social isolation and physical activity. Scoring is done between 0 and 100, with a high score indicating a low QoL.

SECONDARY OUTCOMES:
The Pittsburgh Sleep Quality Index (PSQI) | 15 minutes
  Sleep quality was assessed with the PSQI. The scale consisting of 24 questions in total aims to evaluate the sleep quality of the individual in the last month.PSQI consists of 18 items consisting of 7 components in a 1-month period. These items are scored according to a 4-point Likert scale. PSQI is evaluated over 21 points and a score of 5 and above indicates poor sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Science, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No